CLINICAL TRIAL: NCT04444388
Title: Effect of Cocoa Supplementation in Training Athletes Microbiota and Metabolome: Effects on Acute and Adaptive Exercise
Brief Title: Effect of Cocoa Supplementation in Training Athletes Microbiota and Metabolome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Mar Larrosa, Tenure Professor, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UEM005
Record Dates: First submitted 2020-06-18; First posted 2020-06-23 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Healthy Athletes
MeSH Terms: interventions — Chocolate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cocoa group (Experimental): 5 g/day of flavonoid-rich defatted cocoa for 10 weeks
  Interventions: Dietary Supplement: cocoa
- Placebo group (Placebo Comparator): 5 g/day of maltodextrin for 10 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: cocoa — Sachets of 5 grams of cocoa daily supplementation
  Arms: Cocoa group
Dietary Supplement: Placebo — Sachets of 5 grams of maltodextrin daily supplementation
  Arms: Placebo group

SUMMARY:
It has recently been suggested that cocoa may improve exercise performance and recovery. This study aim to evaluate the plasma and fecal metabolome after 10 weeks of cocoa supplementation during the training period in recreational athletes to detect possible metabolites involved in the observed benefits of cocoa in athletes

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years of age
* high physical condition (VO2 ≥ 55 ml/kg/min)
* BMI 18-25 kg/m2

Exclusion Criteria:

* antibiotics intake during 3 months prior to the study,
* smoking
* nutritional complements
* ergogenic complements
* prebiotics
* probiotics
* vegetarian or vegan diet
* chronic medication
* gastrointestinal surgery
* Any diagnosed disease

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Fecal microbiota | Changes from baseline to 10 weeks of intervention
  Abundance of bacterial taxa determined by 16SRNAr gene sequencing
Fecal metabolome profile | Changes from baseline to 10 weeks of intervention
  Abundance of fecal metabolites, metabolic networks, and metabolic pathways determined by High Pressure Liquid Chromatography-Mass Spectrometry
Plasma metabolome profile | Changes from baseline to 10 weeks of intervention
  Abundance of blood metabolites, metabolic networks, and metabolic pathways activity determined by High Pressure Liquid Chromatography-Mass Spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Mar Larrosa, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Universidad Europea de Madrid, Villaviciosa de Odón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No